CLINICAL TRIAL: NCT00277056
Title: Dysregulated Tyrosine Kinase Signaling in Leukemia
Status: Terminated | Type: Observational
Why Stopped: This is not a clinical trial and was entered in the system in error.
Sponsor: University of New Mexico (Other)
Responsible Party: Sponsor
Other Study IDs: 1602C
Record Dates: First submitted 2006-01-11; First posted 2006-01-13 (Estimated); Last update posted 2024-02-07 (Actual); Status verified 2024-02

CONDITIONS: Leukemia
Keywords: leukemia
MeSH Terms: conditions — Leukemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — blood bone marrow
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Dysregulated Tyrosine Kinase Signaling in Leukemia

DETAILED DESCRIPTION:
Purpose: to look at a number of proteins in the abnormal cells in the blood and/or bone marrow. These proteins make a cell grow or prevent the cell from dying

ELIGIBILITY:
Inclusion Criteria:

* Patients must have newly diagnosed or relapsed leukemia.
* Patients must sign an informed consent.
* Patients will not be excluded if they are receiving chemotherapy.
* Patients with CML, AML, ALL, T/NK leukemia, myelodysplasia, or myeloproliferative disorders will be eligible.
* Patients must be => 18 years of age.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: people with leukemia
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2002-05 (Actual); Primary Completion 2005-10 (Actual); Study Completion 2005-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ian Rabinowitz, MD, Principal Investigator — University of New Mexico
Locations (1):
- University of New Mexico, Albuquerque, New Mexico, United States